CLINICAL TRIAL: NCT04338776
Title: C.L.E.A.R. - Comparing UroLift Experience Against Rezūm
Brief Title: Comparing UroLift Experience Against Rezūm
Acronym: CLEAR
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NeoTract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CP00013
Record Dates: First submitted 2020-04-02; First posted 2020-04-08 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- UroLift (Experimental): Patient randomized to the UroLift arm will receive the FDA-approved UroLift procedure.
  Interventions: Device: UroLift
- Rezūm (Experimental): Patient randomized to the Rezūm arm will receive the FDA-approved Rezūm procedure.
  Interventions: Device: Rezum

INTERVENTIONS:
Device: UroLift — The UroLift System is indicated for the treatment of symptoms due to urinary outflow obstruction secondary to benign prostatic hyperplasia (BPH).
  During the procedure, an implant is delivered into the prostatic lobe obstructing the urethra and restricting urine flow. The distal end of the device is used to compress the lobe then the implant is delivered to retain the lobe in position, thereby increasing the urethral opening and reducing the fluid obstruction through the prostatic urethra.
  Arms: UroLift
Device: Rezum — The Rezūm™ System is intended to relieve symptoms, obstructions, and reduce prostate tissue associated with BPH.
  The Rezūm System is manufactured by Boston Scientific and consists of a radiofrequency (RF) generator and a single-use transurethral delivery device.
  The Rezūm System utilizes radiofrequency current to generate "wet" thermal energy in the form of water vapor, which is then injected into the transition zone and/or median lobe of the prostate tissue in controlled 9-second doses. The vapor that is injected into the prostate tissue rapidly disperses through the interstitial space between the tissue cells. As the vapor cools, it condenses immediately on contact with tissue and the stored thermal energy is released,reducing the volume tissue adjacent to the urethra.
  Arms: Rezūm

SUMMARY:
C.L.E.A.R. Study is poised to compare the patient experience post procedure, including catheterization needs as well as retreatment and BPH medication rates following treatment with either the UroLift® System or Rezūm™ System through 12 months.

DETAILED DESCRIPTION:
Patients will be randomized to either the UroLift or Rezum arm. Post-procedure, subjects who receive a catheter between post-procedure and prior to discharge, will return to office to complete a voiding assessment.

All subjects will be expected to complete questionnaires and assessments, as part of SOC (varies by institution), at day 3, day 7, 2 weeks, 1 month, 3 months and 12 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. Male gender
2. Age ≥ 50 years
3. Diagnosis of symptomatic BPH
4. Prostate volume 30cm3 ≤ 80cm3
5. Willing to sign study informed consent form

Exclusion Criteria:

1. Current urinary tract infection
2. Current catheter dependent urinary retention or PVR >= 500 mL
3. Urethra conditions that may prevent insertion of delivery system into bladder
4. Previous BPH surgical procedure
5. Urinary incontinence presumed due to incompetent sphincter
6. Current gross hematuria
7. Patients with a urinary sphincter implant
8. Patients who have a penile prosthesis
9. Currently enrolled in any other investigational clinical research trial that has not completed the primary endpoint

Min Age: 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must be male. The study is evaluation the population of men diagnosed with benign prostatic hyperplasia.
Enrollment: 120 (Estimated)
Dates: Start 2021-01-22 (Actual); Primary Completion 2025-06-05 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Catheter Independent | Through 1-week
  Number of subjects who are catheter independent and remain catheter independent through 1-week

CONTACTS AND LOCATIONS:
Locations (10):
- United States (7):
  - Tower Urology, Los Angeles, California
  - Comprehensive Urology, Royal Oak, Michigan
  - NYU Winthrop Urology, Garden City, New York
  - Weil Cornell Medical College, Cornell University, New York, New York
  - Urology Austin, Austin, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Urology San Antonio, San Antonio, Texas
- United Kingdom (3):
  - Frimley Park Hospital, Frimley, Camberley
  - NORFOLK and Norwich University Hospital, Norwich, Norfolk
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge